CLINICAL TRIAL: NCT01215539
Title: A SINGLE-ARM, MULTICENTER, PHASE II STUDY OF PANITUMUMAB IN COMBINATION WITH CAPECITABINE / OXALIPLATIN IN FIRST-LINE, WILD-TYPE K-RAS METASTATIC COLORECTAL CANCER PATIENTS.
Brief Title: Study of Panitumumab-Capecitabine-Oxaliplatin In Wild-Type K-Ras Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 6A/09; 2009-012655-26 (EudraCT Number)
Record Dates: First submitted 2010-09-29; First posted 2010-10-06 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab,capecitabine,oxaliplatin (Experimental): Panitumumab will be administered by IV infusion on day 1 of each 3-week cycle prior to the administration of chemotherapy. The starting panitumumab dose is 9 mg/kg.
  Oxaliplatin 130 mg/m2 IV infusion over 2 hours on Day 1 Capecitabine 2000 mg/m2 divided in two doses, orally, on Days 1 - 14
  Interventions: Drug: panitumumab

INTERVENTIONS:
Drug: panitumumab — Panitumumab will be administered by IV infusion on day 1 of each 3-week cycle prior to the administration of chemotherapy. The starting panitumumab dose is 9 mg/kg. Subjects with evidence of complete response, partial response or stable disease will continue to receive the combination of chemotherapy with panitumumab until disease progression, unacceptable toxicity or withdrawal of consent.

SUMMARY:
The purpose of this study is to determine whether panitumumab in combination with capecitabine/oxaliplatin are effective as first-line treatment in wild-type k-ras, metastatic colorectal cancer patients.

DETAILED DESCRIPTION:
This is a single-arm trial in which previously untreated, wild-type k-ras metastatic colorectal cancer patients will receive therapy with the combination of panitumumab with capecitabine and oxaliplatin. During the treatment period of 6 cycles, subjects with evidence of complete response, partial response or stable disease will continue to receive the combination of chemotherapy with panitumumab until disease progression, unacceptable toxicity or withdrawal of consent. Those patients with disease stabilization who are not appropriate for chemotherapy may continue with panitumumab alone. Patients with disease progression will be discontinued from chemotherapy and panitumumab and will be followed every 3 months after the last drug administration until death. Tumor response will be assessed according to the RECIST criteria (investigator's read of scans), every 6 weeks through week 18 and every 3 months thereafter, until disease progression. Disease progression will also be evaluated radiographically at the time of clinical suspicion of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and sign an informed consent
2. Aged 18 years or more
3. Histologically or cytologically-confirmed metastatic adenocarcinoma of the colon and/or rectum
4. Measurable disease according to the RECIST criteria
5. Eastern Cooperative Oncology Group (ECOG) status of 0-2
6. Non-mutated k-ras gene (k-ras status will be assessed by DNA sequencing in codons 12 and 13)
7. Haematologic function: ANC >1.5 x 109/L, Leucocyte count >3000/mm3, Haemoglobin >10g/ d L, PLT >100 x 109/ L
8. Renal function: serum creatinine ≤1.5xUNL or creatinine clearance > 50ml/min
9. Hepatic function:

   * Total bilirubin ≤ 1.5 time the upper normal limit (UNL)
   * ASAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases
   * ALAT ≤ 2.5xUNL in absence of liver metastases, or ≤5xUNL in presence of liver metastases
10. Metabolic function:

    * Magnesium ≥ lower limit of normal.
    * Calcium ≥ lower limit of normal.

Exclusion Criteria:

1. Central nervous system metastases
2. Prior therapy for metastatic disease
3. Adjuvant chemotherapy for the last 6 months
4. Prior anti-EGFR therapy or treatment with EGFR tyrosine kinase inhibitors
5. Prior radiotherapy within 30 days from enrollment
6. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) <=1 year before enrollment
7. History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
8. Inflammatory bowel disease or chronic diarrhea
9. Dihydropyrimidine deficiency
10. Positive test for HIV infection, hepatitis C infection, chronic active hepatitis B infection
11. Any kind of disorder compromising the ability of the patient to give informed consent
12. Any investigational agent within 30 days prior to initiation of the study
13. Any surgical procedure within 28 days prior to initiation of the study
14. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
15. Female subject in childbearing age with a positive pregnancy test at screening or before initiation of study treatment.
16. Subject (male or female) not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Objective Response | Tumor response will be assessed every 6 weeks through week 18 and every 3 months thereafter, until disease progression.
  Response will be evaluated using the RECIST criteria. Response rates will be presented as counts and proportions along with 95% exact confidence intervals.
  An Objective Response is defined as either a Complete Response or a Partial Response. Analysis will be performed in the intent-to-treat population, i.e. all eligible patients enrolled in the study.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  OS will be calculated from the date of enrolment to the date of death or last contact
Progression-Free Survival(PFS) | Tumor response will be assessed every 6 weeks through week 18 and every 3 months thereafter, until disease progression.
  PFS will be calculated from the date of enrolment to the date of disease progression, or death, or last contact. Deaths without a documented progression will be treated as events at the time of death for the PFS analysis.
  Time to event distributions will be estimated using the Kaplan-Meier method.
Adverse Events (AE)of all participants will be recorded and assessed upon signature of the informed consent form, until 30 days after the last administration of study treatment. | 18 months
  Adverse Events will be graded according to the NCI CTCAE v3.0 criteria and will be reported in a frequency table according to the highest severity grade observed per patient
Economic evaluation | 18 months
  The purpose of economic evaluation will be to estimate the total treatment cost of therapy and its componenents from perspective of the health care system and payers. Thus, all resources consumed will be valued to get an idea of the financial implications of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Pectasides, Professor, Study Chair — General Hospital of Athens"Hippokratio", 2nd Dept of Internal Medicine
Locations (12):
- Greece (12):
  - General Hospital of Athens "Hippokratio", 2nd Dept of Internal Medicine, Athens
  - Sotiria General Hospital, 3rd Dept of Medicine, Oncology Unit, Athens
  - General Peripheral Hospital of Athens "Alexandra", Athens
  - Agii Anargiri Cancer Hospital, Oncology Dept, Athens
  - Hygeia Hospital, 2nd Dept of Medical Oncology, Athens
  - Hygeia Hospital, 3rd Dept of Medical Oncology, Athens
  - Metropolitan Hospital, 1st Dept of Medical Oncology, Athens
  - Metropolitan Hospital, 2nd Dept of Medical Oncology, Athens
  - Chania General Hospital, Chania
  - Ioannina University Hospital, Dept of Medical Oncology, Ioannina
  - Rio University Hospital, Dept of Oncology, Pátrai
  - Papageorgiou General Hospital, Dept of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Papaxoinis G, Kotoula V, Giannoulatou E, Koliou GA, Karavasilis V, Lakis S, Koureas A, Bobos M, Chalaralambous E, Daskalaki E, Chatzopoulos K, Tsironis G, Pazarli E, Chrisafi S, Samantas E, Kaklamanos IG, Varthalitis I, Konstantara A, Syrigos KN, Pentheroudakis G, Pectasides D, Fountzilas G. Phase II study of panitumumab combined with capecitabine and oxaliplatin as first-line treatment in metastatic colorectal cancer patients: clinical results including extended tumor genotyping. Med Oncol. 2018 May 31;35(7):101. doi: 10.1007/s12032-018-1160-1. PMID 29855806